CLINICAL TRIAL: NCT05349123
Title: A Home-based Intervention to Promote Mindful Breathing Awareness Through Pursed-lip Breathing Training for COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minnesota HealthSolutions (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mindful Breathing Awareness
Record Dates: First submitted 2022-04-22; First posted 2022-04-27 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Half of the subjects will be randomized to receive home-based PR with the mindful breathing module (intervention group) and half will receive home-based PR (control group).
Who Masked: Outcomes Assessor
Masking Description: Since the patients will know if they have the Pursed Lipped Breathing Application and Spire tags, the outcome assessor will be blinded to which arm received the Application and tags.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Home-based pulmonary rehabilitation that includes health coaching with mindful breathing module
  Interventions: Behavioral: Mindful Breathing; Behavioral: Home-Based Pulmonary Rehabilitation
- Control (Active Comparator): Home-based pulmonary rehabilitation that includes health coaching
  Interventions: Behavioral: Home-Based Pulmonary Rehabilitation

INTERVENTIONS:
Behavioral: Mindful Breathing — Subject will be expected to do 12 weeks of home-based rehabilitation, 6 days a week in their home. The proposed project explores the addition of a mindful breathing module, which involves daily guided breathing practice with feedback to encourage mindful breathing.
  Arms: Intervention
Behavioral: Home-Based Pulmonary Rehabilitation — Subject will be asked to complete exercise guided by a video six days a week and to complete mindful walking six days per week. They will receive weekly health coaching calls.
  Other Names: Health Coaching

SUMMARY:
The Mindful Breathing Laboratory under the direction of Dr. Benzo will complete a randomized controlled trial to evaluate the mindful breathing module. This rigorous study will evaluate home-based PR system compared to the home-based PR system plus mindful breathing module for its effects on breathlessness and emotions. The investigators hypothesize that the intervention will decrease breathlessness while increasing emotional perception, emotional intelligence, and mindfulness.

DETAILED DESCRIPTION:
A total of 50 adults diagnosed with COPD will be enrolled in this study. Half of the subjects will be randomized to receive home-based pulmonary rehabilitation with the mindful breathing module (intervention group) and half will receive home-based pulmonary rehabilitation (control group). Each subject will be consented and trained and then participate in either the intervention or control group. Both groups entail one week of baseline and twelve weeks of home-based pulmonary rehabilitation (health coaching plus activity monitoring). The intervention group will also receive the mindful breathing module during the twelve weeks of home-based pulmonary rehabilitation. The Chronic Respiratory Disease Questionnaire (CRQ) will be administered at baseline, week 12 (after the intervention) and week 24 as the investigators will follow the patients for 3 months after the intervention to document the sustainability of the effects (behavior change).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥40 years old
* Patients must have a diagnosis COPD documented by pulmonary function testing; breathlessness of score 2 or higher by the Medical Research Council Score
* Patients must be a current or previous smoker with at least 10 pack-years of cigarette smoking

Exclusion Criteria:

* Patients with a high likelihood of being lost to follow-up or contact (patients with active chemical dependency), are planning to move out of the state; or are not living in the healthcare area
* Patients with an inability to provide good data or follow commands (patients who are disoriented, have a severe neurologic or psychiatric condition)
* Patients with an inability to do mild exercise (patients who have orthopedic-neurologic problems; patients who have severe heart failure, characterized by an ejection fraction of <20% or by New York Heart Association Class IV disease; patients who should be at complete rest, confined to a bed or chair; or patients in whom any physical activity brings on discomfort and in whom symptoms occur at rest).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 48 | 51
Completed | 48 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 48 | 51 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.551 (6.894) | 70.103 (8.922) | 69.832 (7.957)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 19 | 22 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 45 | 48 | 93
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 47 | 50 | 97
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: Participants]
  Afghanistan | 48 | 51 | 99

OUTCOME MEASURES:

1. Primary Outcome: Breathlessness
Description: Breathlessness as measured by the Chronic Respiratory Disease Questionnaire. The Chronic Respiratory Disease Questionnaire is a 20-question inventory assessing four areas, including dyspnea (breathlessness). Patients rate their experience numerically on a 7-point modified Likert scale of 1 to7 with higher ratings indicating less symptom impairment. Scores are obtained by adding the scores for the items that make up each category and dividing by the number of items. A minimally important difference is a change in score of 0.5 or more.
Time Frame: baseline, 3 months, 6 months
Population: For the Intervention group with mindful breathing module arm, nineteen subjects did not complete the three months or six months questionnaire. Data was not collected or analyzed.
  For the Control group, twenty-six subjects did not complete the three months questionnaire and twenty-eight subjects did not complete the six months questionnaire. Data was not collected or analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 29 | 25
score on a scale
  baseline, 3 months | 0.68 [0.36 to 1.0] | 0.71 [0.19 to 1.22]
  baseline, 6 months | 0.34 [-0.03 to 0.71] | 0.83 [0.11 to 1.55]

2. Primary Outcome: Emotion
Description: Emotion as measured by the Chronic Respiratory Disease Questionnaire. The Chronic Respiratory Disease Questionnaire is a 20-question inventory assessing four areas, including emotion. Patients rate their experience numerically on a 7-point modified Likert scale of 1 to7 with higher ratings indicating less symptom impairment. Scores are obtained by adding the scores for the items that make up each category and dividing by the number of items. A minimally important difference is a change in score of 0.5 or more.
Time Frame: baseline, 3 months, 6 months
Population: For the Intervention group with mindful breathing module arm, nineteen subjects did not complete the three months or six months questionnaire. Data was not collected or analyzed.
  For the Control group, twenty-five subjects did not complete the three months questionnaire and twenty-eight subjects did not complete the six months questionnaire. Data was not collected or analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 29 | 26
score on a scale
  baseline, 3 months | 0.45 [0.01 to 0.88] | 0.55 [0.14 to 0.97]
  baseline, 6 months | 0.35 [0.04 to 0.66] | 0.5 [-0.07 to 1.06]

3. Secondary Outcome: Physical Activity
Description: Physical activity as measured by the ActiGraph, primarily daily steps
Time Frame: baseline, 3 months, 6 months
Population: For the Intervention group with mindful breathing module arm, twenty-one subjects did not complete the three months or six months questionnaire. Data was not collected or analyzed.
  For the Control group, twenty-five subjects did not complete the three months questionnaire and thirty subjects did not complete the six months questionnaire. Data was not collected or analyzed.
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 26
steps per day
  baseline, 3 months | 765.98 [46.16 to 1485.79] | 701.5 [-49.43 to 1452.43]
  baseline, 6 months | -181.78 [-987.65 to 624.09] | 290.36 [-537.44 to 1118.17]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study, approximately six months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/51
Other Adverse Events (participants affected / at risk) | 0/48 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT05349123/Prot_SAP_000.pdf